CLINICAL TRIAL: NCT01498328
Title: A Phase II Study of Rindopepimut/GM-CSF in Patients With Relapsed EGFRvIII-Positive Glioblastoma
Brief Title: A Study of Rindopepimut/GM-CSF in Patients With Relapsed EGFRvIII-Positive Glioblastoma
Acronym: ReACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDX110-06
Expanded Access: NCT03068650 (No longer available)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2017-04

CONDITIONS: Glioblastoma; Small Cell Glioblastoma; Giant Cell Glioblastoma; Gliosarcoma; Glioblastoma With Oligodendroglial Component; Recurrent Glioblastoma; Relapsed Glioblastoma
Keywords: EGFRvIII; Glioblastoma; Rindopepimut; CDX-110; Small cell; Giant cell; Brain Cancer; Brain Tumor; Gliosarcoma; oligodendroglial; radiotherapy; chemoradiation; Tumor; Bevacizumab; Relapsed; Returned; Recurrent; EGFR variant III
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Neoplasms; Recurrence | interventions — Bevacizumab; rindopepimut

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1a: Bevacizumab Naïve with Bevacizumab + rindopepimut. (Experimental): About half of the patients who have never received treatment with bevacizumab will receive rindopepimut/GM-CSF in a blinded fashion in combination with bevacizumab.
  Interventions: Drug: Bevacizumab; Drug: Rindopepimut (CDX-110) with GM-CSF
- Group 1b: Bevacizumab Naïve with Bevacizumab + KLH control (Experimental): About half of the patients who have never received treatment with bevacizumab will receive KLH in a blinded fashion in combination with bevacizumab.
  Interventions: Drug: Bevacizumab; Drug: KLH
- Group 2 and 2C: Refractory to Bevacizumab (Experimental): Patients with progressive disease while currently on or within two months after discontinuing bevacizumab will be administered rindopepimut/GM-CSF while continuing (or restarting if they had stopped bevacizumab).
  Interventions: Drug: Bevacizumab; Drug: Rindopepimut (CDX-110) with GM-CSF

INTERVENTIONS:
Drug: Bevacizumab — A vascular endothelial growth factor (VEGF)-specific humanized monoclonal antibody angiogenesis inhibitor. Infusions of 10 mg/kg of bevacizumab will begin on day 1 and will be administered every two weeks until progression of disease or intolerance during the treatment period.
  Other Names: Avastin
Drug: Rindopepimut (CDX-110) with GM-CSF — Rindopepimut/GM-CSF will initially be given three times, two weeks apart, followed by monthly injections until tumor progression or intolerance. Each dose will be 0.8 mL containing approximately 500 mcg CDX-110 and 150 mcg GM-CSF.
  Arms: Group 1a: Bevacizumab Naïve with Bevacizumab + rindopepimut.; Group 2 and 2C: Refractory to Bevacizumab
Drug: KLH — KLH will initially be given three times, two weeks apart, followed by monthly injections until tumor progression or intolerance. Each dose will be 0.8 mL containing approximately 100 mcg of KLH.
  Arms: Group 1b: Bevacizumab Naïve with Bevacizumab + KLH control

SUMMARY:
The purpose of this research study is to find out whether adding an experimental vaccine called rindopepimut (also known as CDX-110) to the commonly used drug bevacizumab can improve progression free survival (slowing the growth of tumors) of patients with relapsed EGFRvIII positive glioblastoma.

DETAILED DESCRIPTION:
This Phase II study will enroll patients into three groups. Group 1 are patients who have never been treated with bevacizumab. These patients will be randomly assigned to receive either rindopepimut/GM-CSF or KLH, each along with bevacizumab. Treatment assignment for Group 1 will be blinded. Group 2 and Group 2C patients are those who are refractory to bevacizumab (experienced recurrence or progression of glioblastoma while on bevacizumab or within 2 months of discontinuing bevacizumab). These patients will all receive rindopepimut/GM-CSF along with bevacizumab. Patients will be treated until disease progression or intolerance and all patients will be followed for survival. Patients may be treated with other therapies that are not part of the study after discontinuing treatment with the study vaccine.

ELIGIBILITY:
Inclusion Criteria:

Among other criteria, patients must meet the following conditions to be eligible for the study:

1. Age ≥18 years of age.
2. Histologic diagnosis of glioblastoma (WHO Grade IV).
3. Documented EGFRvlll positive tumor status (central lab confirmation).
4. First or second relapse of de novo glioblastoma or first diagnosis or first relapse of secondary glioblastoma.
5. Previous treatment must include surgery, conventional radiation therapy and temozolomide (TMZ).
6. Screening MRI must be obtained at least 4 weeks after any salvage surgery, and at least 12 weeks after radiation therapy.
7. KPS of ≥ 70%.
8. If applicable, systemic corticosteroid therapy must be at a dose of ≤ 4 mg of dexamethasone or equivalent per day during the week prior to Day 1.
9. Evaluable disease in Groups 1 and 2; measurable disease in Group 2C
10. Life expectancy > 12 weeks.
11. Patients in Group 2 and 2C must have had disease progression while receiving bevacizumab or within 2 months of treatment with bevacizumab.

Exclusion Criteria:

Among other criteria, patients who meet the following conditions are NOT eligible for the study:

1. Subjects unable to undergo an MRI with contrast.
2. History, presence, or suspicion of metastatic disease
3. Prior receipt of vaccination against EGFRvIII.
4. Any known contraindications to receipt of study drugs, including known allergy or hypersensitivity to keyhole limpet hemocyanin (KLH), GM-CSF (sargramostim; LEUKINE®), polysorbate 80 or yeast derived products, or a history of anaphylactic reactions to shellfish proteins.
5. Use of non-protein based investigational therapy within 14 days prior to Day 1 or use of antibody-based investigational therapy within 28 days prior to Day 1.
6. Clinically significant increased intracranial pressure (e.g., impending herniation), uncontrolled seizures, or requirement for immediate palliative treatment
7. Evidence of recent hemorrhage on screening MRI of the brain
8. Evidence of current drug or alcohol abuse.
9. Patients in Group 1 must not have received prior treatment with bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-12; Primary Completion 2015-04 (Actual); Study Completion 2016-05-17 (Actual)

PRIMARY OUTCOMES:
Groups 1 and 2: Progression-free survival rate | 6 months post-Day 1
  Evaluate the antitumor activity of rindopepimut in adult patients with relapsed glioblastoma, as measured by the progression-free survival rate at 6 months post-Day 1 (PFS 6).
Group 2C: Objective Response Rate | Every 8 weeks from Day 1 through progression or initiation of other anti-cancer therapy
  Evaluate the anti-tumor activity of rindopepimut in adult patients with relapsed glioblastoma, as measured by the objective response rate (ORR) for patients with measurable disease at study entry.

SECONDARY OUTCOMES:
Safety and Tolerability | Until 28 days or initiation of other anti-cancer treatment, whichever is first
  Safety and tolerability will be evaluated by comparing the treatment regimens in regards to vital sign measurements, physical and neurological examinations, adverse events reporting, and Karnofsky performance status
Anti-tumor activity | During treatment and every 8 weeks through follow up
  Evaluated by comparing the treatment regimens for anti-tumor activity, including objective response rate, overall progression free survival (PFS), and overall survival (OS) for Groups 1 and 2; and PFS6, overall PFS, and OS for Group 2C.
EGFRvIII-specific immune response | Several times during the first month of treatment and then approximately every 8 weeks until treatment is stopped.
  Characterize the EGFRvIII specific immune response to rindopepimut.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center / Barrow Neurological Institute, Phoenix, Arizona
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University of Southern California (USC) Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - University of California San Francisco, San Francisco, California
  - Stanford Cancer Institute, Stanford University, Stanford, California
  - University of Colorado, Denver, Aurora, Colorado
  - Memorial Cancer Institute, Hollywood, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Atlanta Cancer Care, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute and Mass General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Sparrow Cancer Center, Lansing, Michigan
  - John Nasseff Neuroscience Institute, Abbott Northwestern Hospital, 800 e. 28th Str. MR, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New Jersey Neuroscience Institute JFK Medical Center, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Dent Neurologic Institute, 3980 Sheridan Dr, 3rd Flr Clinical Rsch, Amherst, New York
  - The Long Island Brain Tumor Center at Neurology Surgery, P.C., Commack, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - The Preston Robert Tisch Brain Tumor Center; Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Legacy Research Institute, Portland, Oregon
  - Lehigh Valley Hospital-John and Dorothy Morgan Cancer Center, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology Midtown, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - UT Health Science Center, Houston Memorial Hermann Hospital, 6400 Fannin Street, #2800, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Swedish Neuroscience Research, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Reardon DA, Desjardins A, Vredenburgh JJ, O'Rourke DM, Tran DD, Fink KL, Nabors LB, Li G, Bota DA, Lukas RV, Ashby LS, Duic JP, Mrugala MM, Cruickshank S, Vitale L, He Y, Green JA, Yellin MJ, Turner CD, Keler T, Davis TA, Sampson JH; ReACT trial investigators. Rindopepimut with Bevacizumab for Patients with Relapsed EGFRvIII-Expressing Glioblastoma (ReACT): Results of a Double-Blind Randomized Phase II Trial. Clin Cancer Res. 2020 Apr 1;26(7):1586-1594. doi: 10.1158/1078-0432.CCR-18-1140. Epub 2020 Feb 7. PMID 32034072
- [Derived] Gatson NT, Weathers SP, de Groot JF. ReACT Phase II trial: a critical evaluation of the use of rindopepimut plus bevacizumab to treat EGFRvIII-positive recurrent glioblastoma. CNS Oncol. 2016;5(1):11-26. doi: 10.2217/cns.15.38. Epub 2015 Dec 15. PMID 26670466 (Retraction: PMID 26732311 CNS Oncol. 2016;5(2):110)